CLINICAL TRIAL: NCT04629482
Title: The Brain Network Activity of Functional Tasks Performance by Magnetoencephalography for Children
Brief Title: Brain Activity by Magnetoencephalography for Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Professor, Taipei Medical University
Other Study IDs: 2020SKHADR035
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Brain Activity
Keywords: attention deficit hyperactivity disorder; networks; magnetoencephalography; developmental delay; children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with attention deficit hyperactivity disorder with developmental delays: Children with attention deficit hyperactivity disorder with developmental delays
  Interventions: Other: Brain networks activity
- Children with typical development: Children with typical development
  Interventions: Other: Brain networks activity

INTERVENTIONS:
Other: Brain networks activity — The brain network activity under different conditions will be evaluated by magnetoencephalography, including resting, listen to different types of music, watch different types of videos, and interacting with cognitive stimulation conditions.

SUMMARY:
Investigate the differences in activation of brain networks during performing functional tasks for children with attention deficit hyperactivity disorder with developmental delays and typical development

DETAILED DESCRIPTION:
A total of 12 children with attention deficit hyperactivity disorder with developmental delays and12 children with typical development will be enrolled.

The following evaluations will be evaluated by the investigator who is blinded to the group's classification.

Working task-related functions, such as Beery-Buktenica Visual-Motor Integration, Sensory Profile, the Chinese version of Swanson, Nolan and Pelham version IV, and Chinese version of Wechsler Intelligence Scale for Children-IV)

Non-working memory-related functions, such as Pediatric Outcome Data Collection Instrument (PODCI), Child Health Questionnaire- Parent Form (CHQ-PF 28), Pediatric Quality of Life Inventory (PedsQL), and physical function (10 meters normal and fast walking, stair ascent, stair descent, and 5 times chair rising and timed up and go test)

All participants will be investigated by magnetoencephalography and eye-tracking system to identify the difference of brain network activation during resting and performing tasks and between-group differences.

Brain magnetic resonance image study will be performed for matching of brain localization.

ELIGIBILITY:
Inclusion Criteria:

* children with attention deficit hyperactivity disorder with development delays
* intelligence quotient 70 or greater

Exclusion Criteria:

* age less than 4 or greater than 10 of children
* intelligence quotient less than 70

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children diagnosed with attention deficit hyperactivity disorder with developmental delays, aged 4 to 10; and age-sex matched children with typical development
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Brain network activity by magnetoencephalograph | measure simultaneous brain activity by different types of music through study completion, up to 6 minutes
  magnetoencephalography by different types of music
Brain network activity by magnetoencephalography | measure simultaneous brain activity by different types of videos through study completion, up to 10.5 minutes
  magnetoencephalography by different types of videos
Brain network activity by magnetoencephalography | measure simultaneous brain activity by different types of interactive cognitive stimulation through study completion, up to 5 minutes
  magnetoencephalography by different types of interactive cognitive stimulation

OTHER OUTCOMES:
Beery-Buktenica Visual-Motor Integration | before magnetoencephalography examination
  assess visual motor function
Sensory Profile Questionnaire | before magnetoencephalography examination
  assess sensory integration,15 to 85, higher scores mean a better outcome
Swanson, Nolan and Pelham | before magnetoencephalography examination
  assess the symptoms of attention deficit hyperactivity disorders, 0-78, higher scores mean a worse outcome
Wechsler Intelligence Scale for Children | before magnetoencephalography examination
  assess the intelligence, 40-160, higher scores mean a better outcome
Pediatric Outcome Data Collection Instrument | before magnetoencephalography examination
  assess the functional performance, 0-100, higher scores mean a better outcome
Child Health Questionnaire- Parent Form | before magnetoencephalography examination
  assess the family impact, 0-100, higher scores mean a better outcome
Pediatric Quality of Life Inventory | before magnetoencephalography examination
  assess the health-related quality of life, 0-100, higher scores mean a better outcome
10 meters walking speed | before magnetoencephalography examination
  assess normal and fastest walking speed
stairs climbing time | before magnetoencephalography examination
  assess ascent and descent stairs time
chair-rising time | before magnetoencephalography examination
  assess 5 times of chair-rising time
timed up and go | before magnetoencephalography examination
  assess time for stand up from a chair, go around for 3 meters, and sit down to chair

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Ru-Lan, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No